CLINICAL TRIAL: NCT02213796
Title: Population Pharmacokinetics and Monte Carlo Dosing Simulations of Meropenem During the Early Phase of Severe Sepsis and Septic Shock in Critically Ill Patients in Intensive Care Units
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sutep Jaruratanasirikul (Other)
Collaborators: Prince of Songkla University (Other)
Responsible Party: Sponsor-Investigator, Sutep Jaruratanasirikul, Principal investigator, Prince of Songkla University
Organization: Prince of Songkla University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MEROICU14
Record Dates: First submitted 2014-08-08; First posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Initial Phase of Severe Sepsis and Septic Shock
Keywords: meropenem, early phase, severe sepsis and septic shock, critically ill, population pharmacokinetics
MeSH Terms: conditions — Shock, Septic; Sepsis; Critical Illness | interventions — Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1h infusion of 1 g meropenem (Other)
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Meropenem

SUMMARY:
This is a prospective, noncomparative study to assess the pharmacodynamics of meropenem during early phase of severe sepsis and septic shock in critically ill patients in an intensive care unit.

Clinical and laboratory data such as age,sex, body weight, electrolyte, vital signs, APACHE II score, SOFA score, BUN, Cr and blood culture will be collected.

Twelve patients will be enrolled in this study. Meropenem pharmacokinetic will be carried out during the first and second dose after 1g meropenem administration. Blood samples (approximately 3 ml) will be obtained by direct venepuncture at the following time: 0, 0.25, 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 8, 8.5, 9, 9.5, 10, 12, 14 and 16 h.

Meropenem assays will be performed by modified method of Ozkan et al. (Biomed. Chromatogr., 2001).

The pharmacokinetics of meropenem will be modelled from concentration-time profile using compartmental model. Monte Carlo simulation to assess PK/PD index as 40% and 100% T>MIC will be conducted and the results will be reported as % PTA (Probability Target Attainment) and %CFR (Cumulative Faction Response)

DETAILED DESCRIPTION:
Introduction:

Severe sepsis/septic shock are one of the most important reasons for admission the critically-ill patient to Intensive Care Units (ICU) and remaining a major causes of high mortality. Evidently, the fluctuation in pathophysiology, particularly during early phase, of this condition may result in PK alteration and lead to the inadequate antibiotic dosed of standard treatment. Therefore, thearly phase treatment with an appropriate antimicrobial doses that achieved pharmacodynamic target for antimicrobial therapy have been the crucial factor for therapeutic.

Meropenem, a carbapenem antibiotic, is a β-lactam antimicrobial agent with a broad spectrum of activity, coverage of gram-negative bacteria including highly resistant pathogens for instance ESBL-producing or AmpC-mediated b-lactamase producing Enterobacteriaceae. This agent, in common with other β-lactams, is characterized by time-dependent antimicrobial activity, and the exposure time during which the free drug concentrations remains above the minimum inhibitory concentration (T>MIC) is the pharmacokinetic/pharmacodynamic (PK/PD) index that best correlates with efficacy. The majority of previous PK/PDs studies on β-lactams in critically ill patients were mostly conducted in the steady-state period of treatment in which during the early phase of severe sepsis/septic shock was still lacking.

Objectives:

To study the population PK of meropenem and assess the probability of target attainment (PTA) of meropenem inthe initial phases of severe sepsis or septic shock patients in order to be able to optimize dosing recommendations.

Clinical and laboratory data:

Age, sex, body weight, electrolite, vitalsigns, APACHAE II score, BUN, Cr, blood culture

Drug preparation and administration:

The dosage of meropenem was 1-h infusion of 1g diluted in 100 mL of normal saline solution via infusion pump at a constant flow rate every 8 h (q8h) for 16 hours.

Study design:

Prospective non-comparative studyof 9 patients during the initial 24 h of severe sepsis or septic shock. Each subject received a 1-h infusion of 1 g q8h of meropenem for 16 hrs. Monte Carlo simulation were attempted to analyze the pharmacokinetics of experimental data.

Sample collection:

Meropenem PK studies were carried out during the administration of the first and second dose of meropenem (0-16 h after the start of administration of meropenem). Blood samples (ca. 3 mL) were obtained by direct venipuncture at the following times: shortly before (time 0) and then at 0.25, 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 8, 8.5, 9, 9.5, 10, 12, 14 and 16 h after the start of administration of meropenem. All blood samples were added to a heparinized tube, were immediately stored on ice and were centrifuged at 2000 × g at 4◦C for 10 min within 5 min. All plasma samples were stored at -80◦C until analysis within 1 week.

Moropenem assay:

The meropenem assays by method of Ozkan et al. (Biomed Chromatogr, 2001) will be performed at Department of Medicine, Faculty of Medicine.

Duration of study:

Patients will receive a 1-h infusion of 1 g q8h of meropenem for 16 hrs.

Pharmacokinetic and pharmacodynamic analysis:

Concentration of meropenem in plasma will be simulated in Monte Carlo technique to get PK/PD index (40% and 80% PTA)

Sample size: Nine patients with severe sepsis and septic shock.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age > 18 years
2. Patients who diagnosed as severe sepsis or septic shock, either at admission or during the ICU stay. Sepsis is the systemic response to infections defined by two or more of the following conditions: body temperature of >38 oC or <36 oC; heart rate of > 90 beats per min; respiratory rate of >20 breaths per min or a PaCO2 of <32 mmHg; or leucocyte count >12,000 cell/mm3, <4,000 cell/mm3 or 10% immature (band) forms. Severe sepsis is defined by sepsis associated with organ dysfunction, hypoperfusion, or hypotension (systolic arterial pressure <90 mmHg, mean arterial pressure <70 mmHg or a reduction of ≥40 mmHg from baseline). Septic shock is defined by severe sepsis associated with hypotension despite adequate fluid resuscitation

Exclusion Criteria:

1. Patients who are pregnant.
2. Patients who have documented hypersensitivity to carbapenems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Concentration of meropenem in plasma | 16 hour after first dose
  Concentration of meropenem inplasma will be simulated in Monte Carli simulation to assess PK/PD index as 40% and 100 T>MIC and will be reported as %PTA.

CONTACTS AND LOCATIONS:
Overall Officials: Sutep Jaruratanasirikul, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand